CLINICAL TRIAL: NCT07304947
Title: Personalized Cardiac Index-Guided Intraoperative Hemodynamic Management to Improve Postoperative Outcomes in Pediatric Patients With Moyamoya Disease: A Randomized Controlled Trial
Brief Title: Cardiac Index-Guided Intraoperative Hemodynamic Management in Pediatric Moyamoya Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun-hee Kim, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-2411-122-1591
Record Dates: First submitted 2025-11-28; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Moyamoya Disease
MeSH Terms: conditions — Moyamoya Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac index guided hemodynamic management (Experimental)
  Interventions: Procedure: Cardiac Index-Guided Hemodynamic Management
- Blood pressure guided hemodynamic management (Active Comparator)
  Interventions: Procedure: Blood Pressure-Guided Standard Hemodynamic Management

INTERVENTIONS:
Procedure: Cardiac Index-Guided Hemodynamic Management — In the experimental arm, intraoperative hemodynamic management is guided by each patient's baseline cardiac index. Cardiac output is continuously monitored using the LiDCO system after arterial line insertion. Baseline cardiac index is calibrated using transthoracic echocardiography, and intraoperative fluids and vasoactive agents are adjusted to maintain cardiac index within ±20% of baseline. Standard anesthesia monitoring is provided to all patients.
  Arms: Cardiac index guided hemodynamic management
Procedure: Blood Pressure-Guided Standard Hemodynamic Management — In the control arm, intraoperative hemodynamic management follows conventional blood pressure-guided practice. After arterial line placement, the LiDCO device remains connected but the display is concealed during anesthesia. Fluids and vasoactive medications are adjusted according to standard MAP-based management. Standard anesthesia monitoring is provided to all patients.
  Arms: Blood pressure guided hemodynamic management

SUMMARY:
This prospective randomized controlled trial evaluates whether individualized cardiac index-guided intraoperative hemodynamic management reduces postoperative transient ischemic episodes in pediatric patients undergoing encephaloduroarteriosynangiosis (EDAS) for Moyamoya disease. Patients are randomized 1:1 to goal-directed fluid therapy based on baseline cardiac index versus standard arterial pressure-based management. The primary outcome is the incidence of transient ischemic episodes during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients <18 years undergoing EDAS for Moyamoya disease under general anesthesia

Exclusion Criteria:

* ASA physical status 4-5
* Emergency surgery
* Known cardiovascular disease
* Any condition judged inappropriate by investigators

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-12-02 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of transient ischemic episodes during hospitalization | Postoperative hospital stay
  From end of surgery through postoperative hospital discharge, up to 7 days

SECONDARY OUTCOMES:
MRI-confirmed postoperative cerebral infarction | From postoperative Day 0 through Day 7
MRI-confirmed intracranial hemorrhage | From postoperative Day 0 through Day 7
Length of hospital stay | From postoperative Day 0 through Day 7
  Total number of days from the date of surgery to discharge.
Intraoperative fluid volume administered | Intraoperative period
  Total amount of crystalloid and colloid administered during surgery.
Intraoperative vasoactive agent dose | Intraoperative period
  Total dose of vasoactive medications administered during anesthesia.
Intraoperative urine output | Intraoperative period
  Total urine output measured during surgery.
Estimated blood loss | Intraoperative period
  Total estimated blood loss recorded during the surgical procedure.
Duration of anesthesia | Intraoperative period
  Time from induction of anesthesia to completion of anesthesia.
Duration of postoperative mechanical ventilation | From end of surgery until extubation, assessed up to 24 hours
  Total duration of mechanical ventilation following surgery.
Length of ICU stay | From postoperative Day 0 through ICU discharge, assessed up to 14 days
  Number of days spent in the ICU after surgery.
Percentage of anesthesia time with MAP deviating >20% from baseline | Intraoperative period
  Proportion of total anesthesia time during which mean arterial pressure deviates more than 20% from the patient's ward baseline MAP.
Percentage of anesthesia time with cardiac index deviating >20% from baseline | Intraoperative period
  Proportion of total anesthesia time during which cardiac index deviates more than 20% from the patient's baseline cardiac index measured via preoperative echocardiography.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea